CLINICAL TRIAL: NCT02758041
Title: A Study to Evaluate Sebacia Microparticles in Patients With Inflammatory Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sebacia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEB-0294CH, SEB-0400
Record Dates: First submitted 2016-04-19; First posted 2016-05-02 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Facial Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sebacia Microparticles (Experimental)
  Interventions: Device: Sebacia Microparticles

INTERVENTIONS:
Device: Sebacia Microparticles

SUMMARY:
This study is proposed to evaluate Sebacia Microparticle treatment in patients with facial inflammatory acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 16-45 years of age.
2. Moderate to moderately-severe facial inflammatory acne vulgaris
3. Fitzpatrick skin phototype I-III

Exclusion Criteria:

1. Pregnant, lactating, nursing or planning to become pregnant
2. Tattoo in the treatment area
3. Active skin disease, excessive scarring or excess facial hair in the treatment area
4. Certain current or recent acne treatments
5. Recent light treatments including Intense Pulsed Light or other lasers, microdermabrasion or chemical peels in the treatment area
6. Contraindicated for laser treatment, or is unable or unwilling to avoid excessive sun exposure or tanning bed use
7. Known allergy to gold

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Percent reduction in lesion count from baseline | Baseline, Week 12, Week 24, Week 36

SECONDARY OUTCOMES:
Improvement in Investigator Global Acne Score | Baseline, Week 12, Week 24, Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD, PhD, Principal Investigator — Department of Dermatology, Bispebjerg Hospital, Univ of Copenhagen
Locations (3):
- Denmark (2):
  - Lasercenter North, Aalborg
  - Department of Dermatology, Bispebjerg Hospital, Univ of Copenhagen, Copenhagen
- SKINPULSE Dermatology Laser & Beauty Center, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided